CLINICAL TRIAL: NCT05061836
Title: Effect of Using Dextrose-containing Intraoperative Fluid in Children: a Randomized Controlled Trial
Brief Title: Effect of Using Dextrose-containing Intraoperative Fluid in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, patcharee sriswasdi, MD, MPH, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Pediatric Surgery
Keywords: Glucose containing solution; Dextrose containing solution; Dextrose-saline solution; Pediatric fluid; Pediatric hyperglycemia; Pediatric hypoglycemia; Intraoperative glucose; Intraoperative fluid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dextrose0 (Experimental): Acetate Ringer's solution
  Interventions: Drug: Ringer acetate
- Dextrose1 (Experimental): 1.25%dextrose equivalence
  Interventions: Drug: 1.25%Dextrose equivalence
- Dextrose2 (Experimental): 2.5%dextrose equivalence
  Interventions: Drug: 2.5%Dextrose equivalence
- Dextrose5 (Active Comparator): 5%dextrose
  Interventions: Drug: Dextrose 5

INTERVENTIONS:
Drug: Ringer acetate — Patient will receive Acetate Ringer's solution (Acetar) infused at maintenance rate
  Arms: Dextrose0
Drug: 1.25%Dextrose equivalence — 5%dextrose in normal saline (5%DNSS) infused ¼ of maintenance rate
  Arms: Dextrose1
Drug: 2.5%Dextrose equivalence — 5%dextrose in normal saline (5%DNSS) infused ½ of maintenance rate
  Arms: Dextrose2
Drug: Dextrose 5 — 5%dextrose in normal saline (5%DNSS) infused with maintenance rate
  Arms: Dextrose5

SUMMARY:
The glucose-containing fluid was preferred for maintenance fluid in pediatric surgery to prevent hypoglycemic events. This practice can lead to intraoperative hyperglycemia which can induce osmotic diuresis and consequently dehydration and electrolyte disturbances.

As an anesthesiologist, the use of glucose-containing fluid should be reconsidered to avoid these undesirable effects in pediatric surgery.

Our study aims to identify an appropriate use of 5% dextrose containing solution during intraoperative period in children (2 age groups: 1-2 vs 3-5 years old) that can prevent glucose and lipid mobilization without causing hypo/hyperglycemia and provide adequate fluid maintenance in the context of hospitals in Thailand

DETAILED DESCRIPTION:
* In this randomized controlled trial, the investigator will find the difference in pre and postoperative value of base excess among the different fluid groups which is an acid-base parameter indicating volume status and mobilization of lipid stores in each age group (2 age group: 1-2 vs 3-5 years old). Each age group will be divided to:

  1. Group D0: patients will receive Acetate Ringer's solution (Acetar) infused at maintenance rate
  2. Group D1: 5%dextrose in normal saline (5%DNSS) infused ¼ of maintenance rate [resulted in 1.25%dextrose equivalence]
  3. Group D2: 5%DNSS infused ½ of maintenance rate [resulted in 2.5%dextrose equivalence]
  4. Group D5: 5%DNSS infused with maintenance rate
* Patient will be fasting as standard preoperative fasting protocol, and received 5 ml/kg of water at 3 hours prior to surgery
* After standard anesthesia induction and intravenous line (IV) placement, the blood samples will be collected and the POCT glucose will be re-evaluated every 1 hour through the operation to avoid intraoperative hypo/hyperglycemia.
* The first blood sample will be collected after IV line placement and the second blood sample will be collected at the end of surgery. Both blood samples will be sent to the lab to measure blood glucose, serum electrolytes (sodium, potassium, and chloride), acid-base parameters (pH, base excess, standardized bicarbonate, anion gap), endocrine parameters (serum insulin, glucagon, cortisol), and metabolic parameters (free fatty acid, serum ketone, serum lactate).

ELIGIBILITY:
Inclusion Criteria:

1. Children aged of 1 to 5 years
2. ASA physical status 1 and 2
3. Schedule for elective non-abdominal surgery between 1-3 hours under general anesthesia without anticipation of major blood loss at Siriraj Hospital.

Exclusion Criteria:

1. Patients with severe neurologic, cardiac, endocrine, or metabolic disease
2. Patients receiving intravenous fluid preoperatively
3. Patients with history or have known risk of hypoglycemia
4. Patient with severe liver dysfunction

Withdrawal or termination criteria

1. Patients requiring intraoperative blood product transfusion or inotropes infusion
2. Patients who have preoperative hypoglycemia

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The difference in pre and postoperative value of base excess | 1 day
  To find the difference in pre and postoperative value of base excess among the different fluid groups which is an acid-base parameter indicating volume status and mobilization of lipid stores in each age group.

SECONDARY OUTCOMES:
The difference in postoperative value of other acid-base, metabolic, and endocrine parameters | 1 day
  To find the difference in postoperative value of other acid-base, metabolic, and endocrine parameters that indicate mobilization of glucose and lipid stores of each group with different maintenance rate of fluid in each age group and between age group.
Incidence of postoperative base excess value that equal or more negative than -5 of each group | 1 day
  To find the incidence of postoperative base excess value that equal or more negative than -5 of each group with different maintenance rate of fluid in each age group and between age group.
The difference in perioperative blood glucose level among the groups | 1 day
  To find the difference in perioperative blood glucose level among the groups measured during surgery of each group with different maintenance rate of fluid in each age group and between age group.
Incidence of hypotension of each group | 1 day
  To find the incidence of hypotension of each group with different maintenance rate of fluid in each age group and between age group

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nilsson K, Larsson LE, Andreasson S, Ekstrom-Jodal B. Blood-glucose concentrations during anaesthesia in children. Effects of starvation and perioperative fluid therapy. Br J Anaesth. 1984 Apr;56(4):375-9. doi: 10.1093/bja/56.4.375. PMID 6712852
- [Background] Barua K, Rajan S, Paul J, Tosh P, Padmalayan A, Kumar L. Effect of Using Ringer's Lactate, with and without Addition of Dextrose, on Intra-Operative Blood Sugar Levels in Infants Undergoing Facial Cleft Surgeries. Anesth Essays Res. 2018 Apr-Jun;12(2):297-301. doi: 10.4103/aer.AER_53_18. PMID 29962586
- [Background] Suraseranivongse S, Attachoo A, Leelanukrom R, Chareonsawan U, Horatanaruang D. National survey of pediatric anesthesia practice in Thailand. J Med Assoc Thai. 2011 Apr;94(4):450-6. PMID 21591530
- [Background] Sieber FE, Smith DS, Traystman RJ, Wollman H. Glucose: a reevaluation of its intraoperative use. Anesthesiology. 1987 Jul;67(1):72-81. No abstract available. PMID 3111308
- [Background] Lanier WL, Stangland KJ, Scheithauer BW, Milde JH, Michenfelder JD. The effects of dextrose infusion and head position on neurologic outcome after complete cerebral ischemia in primates: examination of a model. Anesthesiology. 1987 Jan;66(1):39-48. doi: 10.1097/00000542-198701000-00008. PMID 3800033
- [Background] Nishina K, Mikawa K, Maekawa N, Asano M, Obara H. Effects of exogenous intravenous glucose on plasma glucose and lipid homeostasis in anesthetized infants. Anesthesiology. 1995 Aug;83(2):258-63. doi: 10.1097/00000542-199508000-00004. PMID 7631946
- [Background] Sumpelmann R, Becke K, Crean P, Johr M, Lonnqvist PA, Strauss JM, Veyckemans F; German Scientific Working Group for Paediatric Anaesthesia. European consensus statement for intraoperative fluid therapy in children. Eur J Anaesthesiol. 2011 Sep;28(9):637-9. doi: 10.1097/EJA.0b013e3283446bb8. PMID 21654319
- [Background] Datta PK, Pawar DK, Baidya DK, Maitra S, Aravindan A, Srinivas M, Lakshmy R, Gupta N, Bajpai M, Bhatnagar V, Agarwala S. Dextrose-containing intraoperative fluid in neonates: a randomized controlled trial. Paediatr Anaesth. 2016 Jun;26(6):599-607. doi: 10.1111/pan.12886. Epub 2016 Apr 16. PMID 27083135
- [Background] HOLLIDAY MA, SEGAR WE. The maintenance need for water in parenteral fluid therapy. Pediatrics. 1957 May;19(5):823-32. No abstract available. PMID 13431307
- [Background] Davis JW, Shackford SR, Mackersie RC, Hoyt DB. Base deficit as a guide to volume resuscitation. J Trauma. 1988 Oct;28(10):1464-7. doi: 10.1097/00005373-198810000-00010. PMID 3172306
- [Background] Beath SV. Hepatic function and physiology in the newborn. Semin Neonatol. 2003 Oct;8(5):337-46. doi: 10.1016/S1084-2756(03)00066-6. PMID 15001122